CLINICAL TRIAL: NCT00542620
Title: A Randomised, Multicentric, Open Labelled, Parallel Group Trial With Insulin Aspart and Insulin Detemir, Investigating the Glycaemic Effect and Profile in Children With Type 1 Diabetes, of Two Separate Levemir® + NovoRapid® Injections and Extemporaneous Mixing - The Paediatric MIXING Trial
Brief Title: Comparison of Insulin Detemir and Insulin Aspart in 2 Separate Injections Twice Daily to Extemporaneous Mixing Injection Regimen Twice Daily - The Paediatric Mixing Trial
Acronym: MIXING
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1813; 2006-006715-77 (EudraCT Number)
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mixed injection (Experimental)
  Interventions: Drug: insulin detemir; Drug: insulin aspart
- Separate injection (Active Comparator)
  Interventions: Drug: insulin detemir; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin detemir — Treat-to-target (individually adjusted) dose titration, s.c. (under the skin) injection, twice a day, mixed with insulin aspart
  Arms: Mixed injection
Drug: insulin aspart — Treat-to-target (individually adjusted) dose titration, s.c. (under the skin) injection, twice a day, mixed with insulin detemir
  Arms: Mixed injection
Drug: insulin detemir — Treat-to-target (individually adjusted) dose titration, s.c. (under the skin) injection, twice a day, injected separately with insulin aspart
  Arms: Separate injection
Drug: insulin aspart — Treat-to-target (individually adjusted) dose titration, s.c. (under the skin) injection, twice a day, injected separately with insulin detemir
  Arms: Separate injection

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to compare two methods of injection in basal-bolus insulin regimen in children with type 1 diabetes with insulin detemir associated with insulin aspart given twice daily in either separate or mixed injections and to investigate if there is any clinical impact in choosing one regimen over another.

ELIGIBILITY:
Inclusion Criteria:

* Parents' Informed Consent (IC) obtained before any trial-related activities
* Obtained child's assent (when possible)
* Type 1 diabetes
* Treatment with insulin detemir and insulin aspart either in extemporaneous mixed or separate injections
* HbA1c (glycosylated haemoglobin A1c) lesser than or equal to 8.6%

Exclusion Criteria:

* History of alcoholism, drug abuse, or psychiatric disease or personality disorders likely to invalidate voluntary consent or to prevent good compliance with the trial protocol
* Mental incapacity, unwillingness or language barrier precluding adequate understanding or co-operation
* Anticipated change or new use in concomitant medication known to interfere with glucose metabolism, such as systemic corticotherapy more than 5 mg/day (prednisone)
* Any other condition that the Investigator (trial physician) feels would interfere with trial participation or evaluation of results

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2007-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Paris, France

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four centres in France
Pre-assignment Details: Children with type 1 diabetes currently treated with insulin detemir and insulin aspart and with a good glycaemic control. At trial entry, subjects must be 6-18 years old with a HbA1c (glycosylated haemoglobin) below or equal to 8.6%
Groups:
- Mixed Injection: Individually adjusted insulin detemir extemporaneous mixed with individually adjusted insulin aspart injected s.c. twice daily (in the morning and in the evening) + extra insulin aspart at lunch and breaks, if needed
- Separate Injection: Individually adjusted insulin detemir and individually adjusted insulin aspart injected separately s.c. twice daily (in the morning and in the evening) + extra insulin aspart at lunch and breaks, if needed
Period: Overall Study
Arm/Group | Mixed Injection | Separate Injection
Started | 13 | 12
Exposed to Drug | 12 (One subject randomly assigned to receive mixed injections, but received a separate injection mode) | 13 (One subject randomly assigned to receive mixed injections, but received a separate injection mode)
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mixed Injection | Separate Injection | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.6 (2.6) | 10.9 (2.5) | 11.3 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  France | 13 | 12 | 25
Diabetes history [Mean (Standard Deviation); unit: years] — Number of years since diagnosis
  years | 6.68 (3.51) | 6.13 (2.38) | 6.42 (2.97)

OUTCOME MEASURES:

1. Primary Outcome: Glycosylated Haemoglobin A1c (HbA1c)
Description: Measured for the Per Protocol (PP) set
Time Frame: Week 0 and Week 8
Population: Per Protocol (PP) analysis set consists of all the ITT (Intention-to-Treat) subjects who did not present any significant protocol deviations that could potentially affect the efficacy results. One subject was excluded from PP as subject received separate injections despite being randomised to receive mixed injections.
Measure: Mean (Standard Deviation); unit: percentage of total haemoglobin
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 12 | 12
percentage of total haemoglobin
  Week 0 | 8.00 (0.54) | 7.77 (0.55)
  Week 8 | 7.63 (0.55) | 8.15 (0.57)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Non-Inferiority or Equivalence — Non-inferiority was considered confirmed if the upper bound of the two-sided 95% confidence interval was below or equal to 0.25% or equivalently if the p-value for the one-sided test of H0: D>0.25% against HA: D=<0.25%, was less than or equal to 2.5%, where D is the mean treatment difference (mixing injections minus separate injections); p = 0.001, ANCOVA — If non-inferiority was confirmed, the superiority of the mixed injection group over separate injection group was to be investigated; Baseline HbA1c as covariate; Median Difference (Final Values) = -0.691, 95% CI [-1.049 to -0.334]

2. Primary Outcome: Glycosylated Haemoglobin A1c (HbA1c)
Description: Measured for the ITT (Intention-to-Treat) set
Time Frame: Week 0 and Week 8
Population: Intention-to-treat (ITT) analysis set consists of all randomised children with a signed informed consent and at least one HbA1c value determined after randomisation. Subjects are analysed based on initial randomisation.
Measure: Mean (Standard Deviation); unit: percentage of total haemoglobin
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 13 | 12
percentage of total haemoglobin
  Week 0 | 7.93 (0.57) | 7.77 (0.55)
  Week 8 | 7.65 (0.53) | 8.15 (0.57)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.003, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Baseline HbA1c as covariate; Mean Difference (Final Values) = -0.594, 95% CI [-0.970 to -0.219]

3. Secondary Outcome: Fructosamine
Time Frame: Week 0 and Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 13 | 12
mmol/L
  Week 0, n=13, 12 | 334.8 (35.9) | 319.8 (22.6)
  Week 8, n=12, 12 | 316.4 (30.1) | 334.8 (41.9)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Superiority or Other; p = 0.573, ANCOVA; With adjustment on baseline fructosamine and the change in insulin administration mode; Mean Difference (Final Values) = -8.35, 95% CI [-38.77 to 22.08], Standard Error of Mean 14.59

4. Secondary Outcome: Self-measured Plasma Glucose Profile (Before Breakfast)
Time Frame: Week 0 and Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 13 | 12
mg/dL
  Week 0 | 190.31 (56.80) | 165.39 (70.28)
  Week 8 | 162.96 (57.46) | 204.75 (59.25)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Superiority or Other; p = 0.063, ANCOVA; With adjustment on baseline value

5. Secondary Outcome: Self-measured Plasma Glucose Profile (After Breakfast)
Time Frame: Week 0 and Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 5 | 7
mg/dL
  Week 0, n=5, 6 | 123.00 (61.9) | 164.89 (73.33)
  Week 8, n=4, 7 | 208.08 (48.19) | 167.98 (70.64)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Superiority or Other; p = 0.389, ANCOVA; With adjustment on baseline value

6. Secondary Outcome: Self-measured Plasma Glucose Profile (Before Dinner)
Time Frame: Week 0 and Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 13 | 12
mg/dL
  Week 0 | 199.14 (42.05) | 201.44 (57.50)
  Week 8 | 185.23 (66.30) | 181.03 (68.41)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Superiority or Other; p = 0.856, ANCOVA; With adjustment on baseline value

7. Secondary Outcome: Self-measured Plasma Glucose Profile (After Dinner)
Time Frame: Week 0 and Week 8
Population: Intention-to-treat (ITT) analysis set consists of all randomised children with a signed informed consent and at least one HbA1c value determined after randomisation. Subjects are analysed based on initial randomisation. CGMS® data not available/sufficient for pre-study evaluation in five subjects or at post-study evaluation in four subjects.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 8 | 6
mg/dL
  Week 0, n=8, 5 | 175.38 (58.47) | 201.80 (59.12)
  Week 8, n=7, 6 | 198.00 (53.85) | 187.67 (85.63)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Superiority or Other; p = 0.917, ANCOVA; With adjustment on baseline value

8. Secondary Outcome: Pharmacokinetics: Cmax of Free Insulin
Description: The observed peak drug concentration at time (T): T0, T0.5hour (hr), T1hr, T1.5hr, T2 hours (hrs), T2.5hrs, T3hrs, T3.5hrs, T4hrs
Time Frame: Week 0 and Week 8
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: pmol/L
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 13 | 12
pmol/L
  Week 0 | 216 (542.4) | 167 (130.4)
  Week 8 | 274 (109.2) | 186 (105.5)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Superiority or Other; p = 0.209, ANCOVA; With adjustment on baseline value

9. Secondary Outcome: Pharmacokinetics: Tmax of Free Insulin
Description: The observed peak drug concentration at time (T): T0, T0.5hour (hr), T1hr, T1.5hr, T2hrs, T2.5hrs, T3hrs, T3.5hrs, T4hrs
Time Frame: Week 0 and Week 8
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: hours
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 13 | 12
hours
  Week 0 | 2.5 (0.74) | 3.0 (0.98)
  Week 8 | 2.5 (0.8) | 1.8 (0.72)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Superiority or Other; p = 0.220, ANCOVA; With adjustment on baseline value

10. Secondary Outcome: Pharmacokinetics: Area Under the Concentration vs. Time Curve From Time Zero to the Time of the Last Measured Level of Free Insulin
Description: as for outcome 9
Time Frame: Week 0 and Week 8
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: pmol.h/L
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 13 | 12
pmol.h/L
  Week 0 | 638.4 (1022.95) | 398.9 (395.19)
  Week 8 | 819.6 (310.41) | 466.2 (266.93)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Superiority or Other; p = 0.234, ANCOVA; With adjustment for baseline value

11. Secondary Outcome: Pharmacokinetics: Area Under the Concentration vs. Time Curve From Time Zero to Infinity of Free Insulin
Description: as for outcome 9
Time Frame: Week 0 and Week 8
Population: as for outcome 7
Measure: Median (Standard Deviation); unit: pmol.h/L
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 11 | 11
pmol.h/L
  Week 0, n=8, 9 | 1441.3 (7516.22) | 752.1 (4128.04)
  Week 8, n=11, 11 | 1981.1 (1442.49) | 672.8 (7156.05)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Superiority or Other; p = 0.534, ANCOVA; With adjustment on baseline value

12. Secondary Outcome: Pharmacokinetics: Terminal Phase Elimination Half-life (T½) - Parameter of Free Insulin
Description: as for outcome 9
Time Frame: Week 0 and Week 8
Population: as for outcome 7
Measure: Median (Standard Deviation); unit: hours
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 11 | 11
hours
  Week 0, n=8, 9 | 3.6 (17.84) | 2.3 (10.93)
  Week 8, n=11, 11 | 2.9 (3.34) | 2.0 (11.62)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Superiority or Other; p = 0.722, ANCOVA; With adjustment on baseline value

13. Secondary Outcome: Pharmacokinetics: Cmax of Insulin Detemir
Description: as for outcome 9
Time Frame: Week 0 and Week 8
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: pmol/L
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 13 | 12
pmol/L
  Week 0 | 10700 (25149.9) | 10500 (6840.2)
  Week 8 | 12000 (23807.2) | 12600 (8426.6)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Superiority or Other; p = 0.727, ANCOVA; With adjustment on baseline value

14. Secondary Outcome: Pharmacokinetics: Tmax of Insulin Detemir
Description: as for outcome 9
Time Frame: Week 0 and Week 8
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: hours
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 13 | 12
hours
  Week 0 | 3.5 (0.93) | 3.5 (0.48)
  Week 8 | 3.5 (0.38) | 3.3 (0.78)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Superiority or Other; p = 0.411, ANCOVA; With adjustment on baseline value

15. Secondary Outcome: Pharmacokinetics: Area Under the Concentration vs. Time Curve From Time Zero to the Time of the Last Measured Level of Insulin Detemir
Description: as for outcome 9
Time Frame: Week 0 and Week 8
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: pmol.h/L
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 13 | 12
pmol.h/L
  Week 0 | 36591.2 (70709.5) | 34653.4 (21243.3)
  Week 8 | 36055.0 (73609.6) | 39757.0 (23076.5)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Superiority or Other; p = 0.471, ANCOVA; With adjustment on baseline value

16. Secondary Outcome: Pharmacokinetics: Area Under the Concentration vs. Time Curve From Time Zero to Infinity of Insulin Detemir
Description: as for outcome 9
Time Frame: Week 0 and Week 8
Population: as for outcome 7
Measure: Median (Standard Deviation); unit: pmol.h/L
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 4 | 6
pmol.h/L
  Week 0, n=4, 3 | 230728.2 (304790.62) | 68509.6 (116350.34)
  Week 8, n=3, 6 | 123555.7 (141207.72) | 362313.5 (4287360.41)

17. Secondary Outcome: Pharmacokinetics: Terminal Phase Elimination Half-life (T½) - Parameter of Insulin Detemir
Description: as for outcome 9
Time Frame: Week 0 and Week 8
Population: Intention-to-treat (ITT) analysis set consists of all randomised children with a signed informed consent and at least one HbA1c value determined after randomisation. CGMS® data not available/sufficient for pre-study evaluation in five subjects or at post-study evaluation in four subjects
Measure: Median (Standard Deviation); unit: hours
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 4 | 6
hours
  Week 0, n=4, 3 | 16.2 (4.12) | 8.2 (6.53)
  Week 8, n=3, 6 | 5.6 (4.2) | 20.8 (249.57)

18. Secondary Outcome: Pharmacokinetics: Cmax of Insulin Aspart
Description: as for outcome 9
Time Frame: Week 0 and Week 8
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: pmol/L
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 13 | 12
pmol/L
  Week 0 | 557 (2784.2) | 762 (378.3)
  Week 8 | 662 (576.3) | 601 (355.3)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Superiority or Other; p = 0.127, ANCOVA; With adjustment on baseline value

19. Secondary Outcome: Pharmacokinetics: Tmax of Insulin Aspart
Description: as for outcome 9
Time Frame: Week 0 and Week 8
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: hours
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 13 | 12
hours
  Week 0 | 2 (0.99) | 2 (0.97)
  Week 8 | 2 (0.53) | 1.5 (0.51)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Superiority or Other; p = 0.1, ANCOVA; With adjustment on baseline value

20. Secondary Outcome: Pharmacokinetics: Area Under the Concentration vs. Time Curve From Time Zero to the Time of the Last Measured Level of Insulin Aspart
Description: as for outcome 9
Time Frame: Week 0 and Week 8
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: pmol.h/L
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 13 | 12
pmol.h/L
  Week 0 | 1546.3 (3163.27) | 1510.9 (963.37)
  Week 8 | 2102.4 (1378.73) | 1540 (894.4)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Superiority or Other; p = 0.166, ANCOVA; With adjustment on baseline value

21. Secondary Outcome: Pharmacokinetics: Area Under the Concentration vs. Time Curve From Time Zero to Infinity of Insulin Aspart
Description: as for outcome 9
Time Frame: Week 0 and Week 8
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: pmol.h/L
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 13 | 12
pmol.h/L
  Week 0, n=10, 11 | 3008.1 (7689.04) | 3006.3 (4458.12)
  Week 8, n=13, 12 | 5674.3 (10668.8) | 3019.9 (1013.19)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Superiority or Other; p = 0.023, ANCOVA; With adjustment on baseline value

22. Secondary Outcome: Pharmacokinetics: Terminal Phase Elimination Half-life (T½) - Parameter of Insulin Aspart
Description: as for outcome 9
Time Frame: Week 0 and Week 8
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: hours
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 13 | 12
hours
  Week 0, n=10, 11 | 2.2 (6.75) | 2 (3.09)
  Week 8, n=13, 12 | 3.5 (41.88) | 1.7 (1.62)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Superiority or Other; p = 0.439, ANCOVA; With adjustment on baseline value

23. Secondary Outcome: Weight Z Score
Description: Z score of weight. To estimate the growth of children, standardised mean weight values were calculated for each month of age and for each sex
Time Frame: Week 0 and Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 13 | 12
Z-score
  Week 0, n=13, 12 | -0.42 (0.71) | 0.19 (0.69)
  Week 8, n=11, 12 | -0.29 (0.65) | 0.26 (0.67)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Superiority or Other; p = 0.202, ANCOVA; With adjustment on baseline value

24. Secondary Outcome: Body Mass Index (BMI) Z Score
Description: Z score of BMI index. To estimate the growth of children, standardised mean BMI values were calculated for each month of age and for each sex
Time Frame: Week 0 and Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 13 | 12
Z-score
  Week 0, n=13, 12 | -0.32 (0.63) | 0.04 (0.86)
  Week 8, n=11, 12 | -0.07 (0.52) | 0.26 (0.73)
Statistical Analysis 1: Comparison: Mixed Injection vs Separate Injection; Test type: Superiority or Other; p = 0.665, ANCOVA; With adjustment on baseline value

25. Secondary Outcome: Incidence of Hypoglycaemic Episodes - All Episodes
Description: Number of hypoglycaemic episodes from Week 0 to Week 8, defined as self-measurement plasma glucose less than 56 mg/dL (3.1 mmol/L). Classified as major, minor or symptoms only. Major if unable to treat her/himself (given the age of the study population, the definition of major hypoglycemia was to be adapted through the investigator's judgment). Minor if able to treat her/himself and plasma glucose below 3.1 mmol/L (56 mg/dL). Symptoms only if able to treat her/himself and no plasma glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L.
Time Frame: Weeks 0-8
Population: All randomised subjects who received at least one treatment dose are taken into account in the safety analysis set. Subjects are analysed based on treatments actually received.
Measure: Number; unit: episodes
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 12 | 13
episodes | 351 | 293

26. Secondary Outcome: Incidence of Hypoglycaemic Episodes - Glycaemia Below 0.56 g/L
Description: Number of minor hypoglycaemic episodes from Week 0 to Week 8, defined as self-measurement plasma glucose below 3.1 mmol/L (56 mg/dL) and the child is able to treat her/himself.
Time Frame: Weeks 0-8
Population: as for outcome 25
Measure: Number; unit: episodes
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 12 | 13
episodes
  With symptoms | 68 | 159
  Without (w/o) symptoms | 75 | 48
  W/o info on presence of symptoms | 23 | 6

27. Secondary Outcome: Incidence of Hypoglycaemic Episodes - Glycaemia Above or Equal to 0.56 g/L
Description: Number of "symptoms only" hypoglycaemic episodes from Week 0 to Week 8, defined as self-measurement plasma glucose higher than or equal to 3.1 mmol/L (56 mg/dL) or no plasma glucose measurement and the child is able to treat her/himself.
Time Frame: Weeks 0-8
Population: as for outcome 25
Measure: Number; unit: episodes
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 12 | 13
episodes
  With symptoms | 49 | 46
  Without (w/o) symptoms | 131 | 33
  W/o information on presence of symptoms | 5 | 1

28. Secondary Outcome: Percentage of Children Assessing Insulin Therapy Injection Pain as "Sad Face"
Description: Via a paper diary, the children perceived insulin therapy injection pain by using a four-grade facial visual analogue scale (VAS): very sad face, sad face, happy face or very happy face.
Time Frame: Week 0 and Week 8
Population: as for outcome 25
Measure: Number; unit: percentage of subjects
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 12 | 13
percentage of subjects
  Week 0 | 45 | 33
  Week 8 | 0 | 23

29. Secondary Outcome: Percentage of Children Assessing Insulin Therapy Injection Pain as "Happy Face"
Description: as for outcome 28
Time Frame: Week 0 and week 8
Population: as for outcome 25
Measure: Number; unit: percentage of subjects
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 12 | 13
percentage of subjects
  Week 0 | 27 | 50
  Week 8 | 81 | 69

30. Secondary Outcome: Percentage of Children Assessing Insulin Therapy Injection Pain as "Very Happy Face"
Description: as for outcome 28
Time Frame: Week 0 and Week 8
Population: as for outcome 25
Measure: Number; unit: percentage of subjects
Arm/Group | Mixed Injection | Separate Injection
Number analyzed (Participants) | 12 | 13
percentage of subjects
  Week 0 | 27.3 | 16.7
  Week 8 | 18.2 | 7.7

ADVERSE EVENTS:
Time Frame: Adverse events are collected during treatment period (8 weeks)
Description: All randomised subjects who received at least one treatment dose are taken into account in the safety analysis set. Subnjects are analysed based on treatments actually received.
Arm/Group | Mixed Injection | Separate Injection
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 5/12 | 9/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mixed Injection (N=12) | Separate Injection (N=13)
Rhinitis (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Enterobiasis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Orthodontic procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Steering Committee has the right to publish the entire results of the trial. Any such scientific paper, presentation, communication, or other information concerning the investigation must be approved by the Steering Committee, and copies submitted in writing to Novo Nordisk prior to submission for publication/presentation for comments. Comments will be given within four weeks from receipt of the manuscript.